CLINICAL TRIAL: NCT05733195
Title: The Study of Biomarker in Early Diagnosis of Gestational Diabetes Mellitus by Metabolomics
Brief Title: The Study of Biomarker in Early Diagnosis of GDM by Metabolomics
Acronym: GDM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-3582
Record Dates: First submitted 2022-12-26; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes Mellitus; Metabolomics Detection; Biomarker in Early Diagnosis
Keywords: GDM; Metabolomics detection; Biomarker in Early Diagnosis
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with GDM: All basic information was collected in the first trimester, and all subjects underwent OGTT (75g glucose) at 24-28 weeks of gestation. GDM will be diagnosed using the criteria of the IADPSG. At four time points during pregnancy (6-13 weeks, 24-28 weeks, 36-weeks before delivery, and 6 weeks after delivery), blood samples of 5ml were collected from each subject at each time point without increasing the number of blood samples. In the GDM group, blood samples were collected at the same time during routine visit 6 weeks after delivery. The relevant broad metabolomics and targeted vitamin profiles were also detected.
  Interventions: Other: OGTT test
- Women with no-GDM: All basic information was collected in the first trimester, and all subjects underwent OGTT (75g glucose) at 24-28 weeks of gestation. GDM will be diagnosed using the criteria of the IADPSG. At three time points during pregnancy (6-13 weeks, 24-28 weeks, 36-weeks before delivery), blood samples of 5ml were collected from each subject at each time point without increasing the number of blood samples. The relevant broad metabolomics and targeted vitamin profiles were also detected.
  Interventions: Other: OGTT test

INTERVENTIONS:
Other: OGTT test — The OGTT test (75g glucose) was performed between 24 and 28 weeks of gestation. GDM will be diagnosed using the criteria of the IADPSG.

SUMMARY:
Gestational Diabetes Mellitus (GDM) refers to abnormal glucose metabolism during pregnancy, in which elevated blood glucose is first found during pregnancy and meets the criteria for diabetes. In recent years, with the increase of obese women of childbearing age, the incidence of GDM has been rising, the current global average incidence is about 14%, and the incidence in China has increased from 2% in 1999 to 5%-8% at present. If one-step diagnosis is used, the rate will be between 13%-17%, which will greatly increase the social burden. Gestational diabetes mellitus (GDM) significantly increases the risk of diseases for pregnant women and infants, such as abortion and premature delivery, concurrent hypertension, concurrent infection, metabolic disorders, postpartum diabetes, macrosomia, fetal malformation, neonatal hypoglycemia, neonatal respiratory distress syndrome, and so on. It is one of the important public health problems threatening human health. Therefore, the accurate diagnosis of GDM is of great clinical significance for the timely formulation of intervention and treatment measures, reducing the risk of maternal and infant diseases and improving the level of public health.

DETAILED DESCRIPTION:
The study will follow a prospective cohort design and be conducted in Peking Union Medical College Hospital. All basic information was collected in the first trimester, and all subjects underwent OGTT (75g glucose) at 24-28 weeks of gestation. GDM will be diagnosed using the criteria of the IADPSG. At four time points during pregnancy (6-13 weeks, 24-28 weeks, 36-weeks before delivery, and 6 weeks after delivery), blood samples of 5ml were collected from each subject at each time point without increasing the number of blood samples. In the GDM group, blood samples were collected at the same time during routine visit 6 weeks after delivery. The relevant broad metabolomics and targeted vitamin profiles were also detected. Meanwhile, blood glucose values at the corresponding time points were collected. Using these variables, we will combine the metabolomics information to screen a predictive marker for GDM in Chinese reproductive age population.

ELIGIBILITY:
Inclusion Criteria:

* First trimester (6-13 weeks)；Pregnant women with a singleton pregnancy；Pregnant women who are registered at the hospital and have regular antenatal check-ups；Pregnant women who volunteered for the study were required to sign an informed consent form

Exclusion Criteria:

* Pregnant women with known type 1 or type 2 diabetes mellitus；Pregnant women with hyperlipidemia and hyperbilirubinemia；Pregnant women with hepatic and renal insufficiency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnancies with gestational diabetes mellitus and no gestational diabetes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
GDM（Pregnancies with gestational diabetes mellitus and no gestational diabetes） | 24-28weeks
  For pregnant women without diabetes before pregnancy, 75g glucose tolerance test (OGTT) was performed at 24-28 weeks of pregnancy as a diagnostic test. The cutting value was that the blood glucose level reached or exceeded 5.1mmol/L, 10.0mmol/L and 8.5mmol/L 0、 1 and 2 hours after taking sugar, respectively. Using standard of the International Association of Diabetes and Pregnancy Study Group (IADPSG), GDM is diagnosed with blood glucose at any point or above the above values.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No